CLINICAL TRIAL: NCT03838419
Title: Intraoperative Electron Radiotherapy for Low-risk Early Breast Cancer
Acronym: COSMOPOLITAN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Juergen Debus, Principal Investigator, University Hospital Heidelberg
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: COSMOPOLITAN
Record Dates: First submitted 2019-02-08; First posted 2019-02-12 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BCS + WBI (Active Comparator): breast conserving surgery followed by whole breast irradiation
  Interventions: Radiation: whole breast irradiation
- BCS + IORT (Experimental): Breast conserving surgery incl intraoperative radiotherapy
  Interventions: Radiation: intraoperative radiotherapy

INTERVENTIONS:
Radiation: intraoperative radiotherapy — IORT with 21 Gy prescribed to the 90% isodose line
  Other Names: IORT
  Arms: BCS + IORT
Radiation: whole breast irradiation — hypofractionated WBI Total dose 40.05 Gy (15 x 2.67 Gy)
  Other Names: WBI
  Arms: BCS + WBI

SUMMARY:
Breast cancer is the most frequent malignancy in women. Standard therapy for early-stage breast cancer is breast conserving surgery (BCS) followed by adjuvant whole breast irradiation (WBI), which usually requires a treatment time of 3-6 weeks. Several randomized controlled trials (RCTs) demonstrated that postoperative WBI after BCS significantly decreased the risk of local (in-breast) recurrence and improved breast cancer mortality as well as survival. However, one of the most common side-effects of radiotherapy is fatigue, which is reported in up to 80% of cancer patients during treatment. Especially in early-stage breast cancer patients it might be the only serious side-effect following adjuvant irradiation, as fatigue often significantly reduces quality of life due to resulting functional impairment and psychological distress. Fatigue additionally has a distinct socioeconomic impact: 75% of patients and 40% of caregivers are forced to change their employment status due to cancer-related fatigue.

For reducing treatment-related toxicity, several RCTs consequently addressed the question whether adjuvant WBI could be omitted in early-stage, low risk breast cancer patients treated with endocrine therapy. However, all these trials detected up to seven-time increased local recurrence rates without WBI following BCS. Both, longer duration of radiotherapy and larger radiation field sizes are known to be associated with increase in treatment-related fatigue. Accelerated partial breast irradiation (APBI), delivered exclusively to the original tumor location and not to the surrounding breast tissue, might therefore be an alternative treatment option with fewer side-effects for early-stage, low risk breast cancer patients. Few previous trials have already reported comparable outcomes for highly selected low-risk breast cancer patients for APBI compared to conventional WBI. First results also point out that APBI compared to WBI might be associated with less severity and intensity of fatigue.

One method for APBI is single-dose intraoperative radiotherapy (IORT) delivered directly to the tumor after resection. Data is still limited for APBI, hence current international and German guidelines suggest the use of APBI for low-risk early stage breast cancer patients but recommend the application of APBI preferably within a clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed invasive breast cancer
* Total tumor size < 2.5 cm
* cN0
* estrogen receptor positive, HER2-receptor negative on immunohistochemistry
* age >= 50 years
* ECOG (Eastern Cooperative Oncology Group) Performance status ≤ 2
* Ability of subject to understand character and individual consequences of the clinical trial
* Written informed consent (must be available before enrolment in the trial)

Exclusion Criteria:

* G3
* Extensive microcalcifications
* Invasive lobular carcinoma
* Clinically involved lymph nodes
* No invasive axillary lymph node staging planned
* Patients with significant mental or physical comorbidities that preclude regular follow-up
* Neoadjuvant chemotherapy or neoadjuvant endocrine therapy
* previous radiotherapy of the breast
* Known carcinoma < 5 years ago (excluding Carcinoma in situ of the cervix, basal cell carcinoma, squamous cell carcinoma of the skin) requiring immediate treatment interfering with study therapy
* Pregnant or lactating women
* Participation in another competing clinical study or observation period of competing trials

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2030-05-01 (Estimated)

PRIMARY OUTCOMES:
Fatigue 12 weeks | 12 weeks
  Assessment of fatigue from baseline (before treatment start) compared to 12 weeks after treatment start as assessed by the FACIT (Functional Assessment of Cancer Therapy) Fatigue Assessment Questionnaire. Scale ranges from 0 (no fatigue) to 52 (maximum fatigue).

SECONDARY OUTCOMES:
Fatigue 5 weeks, 6 months, 2 years, 5 years after treatment start | 5 weeks, 6 months, 2 years, 5 years after treatment start
  Assessment of fatigue from baseline (before treatment start) compared to 5 weeks, 6 months, 2 years, 5 years after treatment start as assessed by the FACIT Fatigue. Scale ranges from 0 (no fatigue) to 52 (maximum fatigue).Assessment Questionnaire.
Local tumor control in the index quadrant of the breast | 2 years and 5 years after treatment start
  Local tumor control in the index quadrant of the ipsilateral breast as a secondary endpoint is defined as no tumor relapse in the breast tissue quadrant of the initial tumor/ at the site of surgical intervention. Local tumor control in the index quadrant of the ipsilateral breast is used as an additional secondary endpoint to distinguish between true local recurrences in the index quadrant from second (or new) ipsilateral carcinomas in other quadrants. In the intraoperative study arm (arm B) only the former tumor bed is irradiated, while in study arm A the whole breast tissue is irradiated.
  Local tumor control in the index quadrant of the breast is taken as number of days from randomization until local tumor progression, death without prior local progression, or end of follow-up. For patients alive and not diagnosed with local progression at the end of the study, the local control time will be censored at the time of the last study visit.
Local tumor control in the ipsilateral breast | 2 years and 5 years after treatment start
  Local tumor control in the ipsilateral breast as a secondary endpoint is defined as no tumor relapse in the whole ipsilateral breast tissue. Local tumor control in the ipsilateral breast is taken as number of days from randomization until local tumor progression, death without prior local progression, or end of follow-up. For patients alive and not diagnosed with local progression at the end of the study, the local control time will be censored at the time of the last study visit.
  Local tumor control in the index quadrant of the breast is taken as number of days from randomization until local tumor progression, death without prior local progression, or end of follow-up. For patients alive and not diagnosed with local progression at the end of the study, the local control time will be censored at the time of the last study visit.
Quality of life employing EORTC (European Organisation for Research and Treatment of Cancer) Quality of life questionnaires (QLQ)-C30 | 5 weeks, 12 weeks, 6 months, 2 years, 5 years after treatment start
  QoL will be analyzed with the help of the EORTC QLQ-C30. Scores are interpreted according to the guidelines of the EORTC Scoring Manual.
Quality of life employing BREAST-Q questionnaire | 5 weeks, 12 weeks, 6 months, 2 years, 5 years after treatment start
  The BREAST-Q questionnaire is specifically designed for patients undergoing BCS measuring quality-of-life (QOL) and satisfaction. Patients are asked to rate each item question on a four-point scale. The BREAST-Q is separated into a pre- and post-surgery version.
Quality of life employing BCTOS (Breast Cancer Treatment Outcome Scale) questionnaire | 5 weeks, 12 weeks, 6 months, 2 years, 5 years after treatment start
  The Breast Cancer Treatment outcome scale (BCTOS-12) contains 12 items, which are assigned to two internally consistent subscales: 1) Functional Status, 2) Aesthetic Status. Patients are instructed to rate each item of the BCTOS-12 on a four-point scale evaluating the differences between the treated and the untreated breast (1 = no difference, 4 = large difference). The score for each subscale is the mean of the ratings over all items belonging to that subscale. A higher score reflects a poorer status (i.e. a larger difference between the treated and the untreated breast).
distant tumor control | 2 years and 5 years after treatment start
  Distant tumor control is defined as no occurrence of distant metastases (lymph node metastases in the axilla, supraclavicular fossa and internal mammary chain are not classified as distant metastases, see above). Distant tumor control is defined as number of days from randomization until occurrence of distant metastases, death without prior distant progression, or end of follow-up. For patients alive and not diagnosed with distant progression at the end of the study, the distant tumor control time will be censored at the time of the last study visit.
Overall survival | 2 years and 5 years after treatment start
  Overall survival time, defined as number of days from randomization until death or end of follow-up. For patients alive at the end of the study, the overall survival time will be censored at the time of the last visit or follow-up contact.
Disease-free survival | 2 years and 5 years after treatment start
  Disease-free survival, defined as number of days from randomization until the first occurrence of local recurrence, regional lymph node metastases, distant metastases, tumor-related death, death without prior progression, or end of follow-up. For patients alive and not diagnosed with progression at the end of the study, the disease-free survival time will be censored at the time the patient was last known to be free of progression of tumor disease.
Secondary malignancies | 2 years and 5 years after treatment start
  Frequency of secondary malignancies after 2 and 5 years will be assessed
Acute toxicity | 5 weeks after treatment start
  Detailed acute potentially therapy-related toxicity will be assessed during each follow-up visit and documentation of side-effects with Common Terminology Criteria for Adverse Events and with the Radiation Therapy Oncology Group (RTOG)/ European Organization for Research and Treatment of Cancer (EORTC) Late Radiation Morbidity Scoring System Schema. Documentation of toxicity will mainly focus on breast shrinkage/distortion, breast induration/ fibrosis, change of skin appearance, telangiectasia, breast oedema, numbness, fat necrosis and local pain.
Chronic toxicity | 6 months, 2 years and 5 years after treatment start
  Detailed chronic potentially therapy-related toxicity will be assessed during each follow-up visit and documentation of side-effects with Common Terminology Criteria for Adverse Events and with the Radiation Therapy Oncology Group (RTOG)/ European Organization for Research and Treatment of Cancer (EORTC) Late Radiation Morbidity Scoring System Schema. Documentation of toxicity will mainly focus on breast shrinkage/distortion, breast induration/ fibrosis, change of skin appearance, telangiectasia, breast oedema, numbness, fat necrosis and local pain.
Cosmesis | 5 weeks, 12 weeks, 2 years, 5 years after treatment start
  Photographic assessments before and after BCS will be taken at baseline and during follow up visits. Evaluation of breast cosmesis will be performed according to the proposed method by Vrieling et al (Schmidt ME, Chang-Claude J, Vrieling A, et al. Fatigue and quality of life in breast cancer survivors: temporal courses and long-term pattern. Journal of cancer survivorship : research and practice 2012;6:11-19.)
Regional tumor control | 2 years and 5 years after treatment start
  Regional tumor control is regarded as no occurrence of regional lymph node metastases (axilla, supraclavicular fossa, internal mammary chain). Regional tumor control is defined as number of days from randomization until occurrence of regional lymph node metastases, death without prior regional tumor progression, or end of follow-up. For patients alive and not diagnosed with regional progression at the end of the study, the regional tumor control time will be censored at the time of the last study visit.

OTHER OUTCOMES:
Explorative Endpoint | after surgery
  Gene expression analysis using the Prosigna/ PAM (Prediction-Analysis-of-Microarray) 50-assay The Prosigna/PAM50-assay will be applied on the operatively resected tumor tissue according to manufactor's instructions

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Heidelberg, Radiation Oncology, Heidelberg, Germany

REFERENCES:
- [Derived] Forster T, Jakel C, Akbaba S, Krug D, Krempien R, Uhl M, Hafner MF, Konig L, Koerber SA, Harrabi S, Bernhardt D, Behnisch R, Krisam J, Hennigs A, Sohn C, Heil J, Debus J, Horner-Rieber J. Fatigue following radiotherapy of low-risk early breast cancer - a randomized controlled trial of intraoperative electron radiotherapy versus standard hypofractionated whole-breast radiotherapy: the COSMOPOLITAN trial (NCT03838419). Radiat Oncol. 2020 Jun 1;15(1):134. doi: 10.1186/s13014-020-01581-9. PMID 32487184